CLINICAL TRIAL: NCT06066216
Title: Efficacy and Safety of Cadonilimab (AK104) Plus Chemotherapy in the Treatment of Recurrent or Advanced Endometrial Cancer: a Multicenter, Prospective Phase II Trial
Brief Title: Cadonilimab (AK104) Plus Chemotherapy in Patients With Recurrent or Advanced Endometrial Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Collaborators: Fujian Provincial Hospital (Other); The First Affiliated Hospital of Nanchang University (Other); Zhangzhou Affiliated Hospital of Fujian Medical University (Other); The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-C-M-0032
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-10

CONDITIONS: Endometrial Cancer; Endometrial Adenocarcinoma
Keywords: Endometrial Cancer; Immune Checkpoint Inhibitors (ICIs); Anti-PD-1/CTLA4 bi-specific antibody; Antiangiogenic agents; Chemotherapy
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Carboplatin; Cisplatin; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab+carboplatin/cisplatin+paclitaxel (Experimental): Cadonilimab (10 mg/kg, administered on the first day of each cycle, Q3W, until there is no clinical benefit)+ carboplatin(AUC=4-5, d1, Q3W, 6cycles) or cisplatin(75 mg/m2, d1, Q3W, 6cycles), +Paclitaxel(175 mg/m2, d1, Q3W, 6cycles), every 3 weeks (21 days) is a treatment cycle
  Interventions: Drug: Cadonilimab; Drug: Carboplatin; Drug: Cisplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Cadonilimab — Injectable solution
  Other Names: AK104
Drug: Carboplatin — Injectable solution
Drug: Cisplatin — Injectable solution
Drug: Paclitaxel — Injectable solutionS

SUMMARY:
This is an open-label, multi-center Phase II study of cadonilimab (AK104) combined with chemotherapy in patients with recurrent or advanced endometrial cancer. The primary objective is to evaluate objective response rate of cadonilimab plus chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patients must have had measurable stage III,IVA or recurrent endometrial cancer,and not suitable for curative radiotherapy or surgery.
3. All patients were required to have histologic confirmation of the original primary tumor (submission of pathology report(s) is required). Patients with the following histologic types were eligible: Endometrioid adenocarcinoma, serous adenocarcinoma, mucinous adenocarcinoma, dedifferentiated/undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, carcinosarcoma, etc.
4. The subject has not received systematic chemotherapy in the advanced or recurrent disease, but is allowed to receive neoadjuvant therapy, adjuvant therapy (including chemotherapy, radiotherapy, or endocrine therapy) in the initial treatment stage, and the last adjuvant chemotherapy is required to be completed at least 6 months before enrollment. The final adjuvant radiotherapy, palliative radiotherapy (such as radiotherapy for bone metastases), and endocrine therapy should be completed at least 3 weeks before enrollment. For palliative radiotherapy of central nervous system (CNS) diseases, washout is allowed for one week.
5. Recurrent endometrial cancer or advanced endometrial cancer that are not suitable for local treatment (including those with extensive abdominal and pelvic lesions, distant metastases, and those who cannot tolerate radiotherapy or surgery, if it is estimated that patients who may achieve surgery or radiotherapy after treatment are not suitable for enrollment).
6. Prior antiangiogenic therapy is permitted.
7. Signed Informed Consent Form (ICF).
8. Provide tumor tissue samples fixed in formalin and embedded in paraffin for pathological examination
9. In patients with measurable disease, lesions are defined and monitored by RECIST v1.1.
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
11. Has adequate organ function as defined by the following criteria:

1) Blood routine examination standards to meet: (no blood transfusion within 14 days)：

* Hemoglobin of ≥90 g/L, white blood cell (WBC) ≥3×109/L, absolute neutrophil count (ANC) ≥1.5×109/L, platelets ≥100 ×109/L 2) Biochemical examination should meet the following criteria：
* Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 × ULN (however, patients with known liver metastasis who have AST or ALT level ≤ 5 × ULN may be enrolled)
* Serum creatinine ≤ 1.5 × ULN 3) Urine protein ≤(++) , or 24-hour urine protein quantification less than 1 g; 4) International standard ratio (INR) and activated partial thromboplastin time ≤1.5 uln (unless anticoagulant therapy is used because of disease) ; 12. Adverse events from any previous treatment, except for symptomatic stable sensory neuropathy or alopecia ≤ CTCAE Grade 2, have returned to ≤ CTCAE grade 1 or baseline, except anemia; 13. Women of childbearing potential should have a negative serum or urine pregnancy test prior to receiving the first dose of study treatment; and should be willing to use one acceptable contraception (i.e., oral contraceptives, condoms, intrauterine devices [IUDs]) throughout the period of taking study treatment and for at least 3 months after the last dose of study drug(s).

  14. Life expectancy exceeds 3 months.

Exclusion Criteria:

1. Other malignant tumors in the past (within 5 years) or at the same time, excluding cured local tumors (such as basal cell skin cancer, squamous cell skin cancer, superficial bladder cancer, cervical carcinoma in situ, breast carcinoma in situ, etc.) and breast cancer and thyroid cancer that have no recurrence more than 3 years after the completion of radical surgery.
2. Had received immunotherapy in the past, it includes immune checkpoint inhibitors (such as anti-PD-1 antibody, anti-PD-L1 antibody, anti-CTLA-4 antibody, etc.) , immune checkpoint agonists (such as ICOS, CD40, CD137, GITR, OX40 antibody, etc.) , immune cell therapy, etc. Such subjects may be admitted with the consent of the sponsor.
3. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
4. Previous history of immunodeficiency; HIV antibody positive; Current long-term use of systemic corticosteroids or other immunosuppressants
5. Subjects who are known to have active pulmonary tuberculosis (TB) and are suspected to have active TB need to undergo clinical examination to exclude them; Known active syphilis infection.
6. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
7. Previous history of non-infectious pneumonia/interstitial lung disease requiring systemic glucocorticoid treatment or current presence of non-infectious pneumonia.
8. Serious infections occur within 4 weeks before the first administration, including but not limited to comorbidities, sepsis, or severe pneumonia that require hospitalization; Active infections (excluding antiviral treatment for hepatitis B or C) that have received systemic anti-infective treatment within two weeks prior to the first administration.
9. Untreated subjects with active hepatitis B (HBSAg positive and HBV-DNA above 1000 copies/ml (200 IU/ml) or above the lower limit of detection, whichever is higher), for subjects with Hepatitis B, anti-HBV therapy was required during study treatment; subjects with active hepatitis C (HCV antibody positive and HCV-RNA levels above the lower limit of detection) .
10. Those who had a major surgical procedure or major trauma within 30 days before the first dose, or who had a major surgical plan within 30 days after the first dose (at the investigator's discretion); Minor local procedures (excluding central venous catheterization via peripheral venipuncture and implantable venous accessport) were performed within 3 days before the first dose.
11. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.
12. There are currently uncontrolled comorbidities, including but not limited to symptomatic congestive heart failure (grade 2 and above according to the New York Heart Association functional classification), unstable angina, acute myocardial ischemia, poorly controlled arrhythmia, decompensated liver cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders, severe active peptic ulcer disease or gastritis, Mental illness/social status that may limit subjects' compliance with research requirements or affect their ability to provide written informed consent.
13. Previous history of myocarditis, cardiomyopathy, and malignant arrhythmia. Unstable angina, myocardial infarction, congestive heart failure, or vascular disease requiring hospitalization (such as aortic aneurysm at risk of rupture), or other cardiac impairment (such as poorly controlled arrhythmias, myocardial ischemia) that may affect study drug safety evaluation within 12 months prior to first administration of study drug; A history of esophageal Gastric varices, severe ulcers, unhealed wounds, gastrointestinal perforation, abdominal fistula, tumor-related gastrointestinal obstruction, intra-abdominal abscess, or acute gastrointestinal bleeding in the 6 months before the first dose; Any arterial thromboembolic event, NCI CTCAE version 5.0 Grade 3 or higher, venous thromboembolism, transient cerebral ischemia, cerebrovascular accident, Hypertensive crisis, or hypertensive encephalopathy, occurred within 6 months before the first dose; Acute exacerbation of chronic obstructive pulmonary disease within 1 month of first dose
14. A history of incurable abdominal fistula or gastrointestinal perforation; During the screening period, imaging revealed obvious tumor invasion of the intestinal wall.
15. During screening, imaging or clinical findings of gastrointestinal obstruction, including incomplete obstruction.
16. Previous history of severe bleeding or coagulation disorders; during screening, imaging showed that the neoplasm surrounded major blood vessels or had obvious necrosis and cavitation, and the investigators believed that participation in the study might increase risk of bleeding.
17. Toxicities from previous antitumour therapy did not resolve, defined as toxicities that did not return to grade 0 or 1 of NCI CTCAE version 5.0, or levels specified in the inclusion/exclusion criteria; Except for alopecia and sequelae of neurotoxicity related to previous platinum therapy. For subjects who experienced irreversible toxicity and are expected to not worsen after the administration of the study drug (such as hearing loss), as well as subjects who have long-term toxicity caused by radiotherapy and cannot be restored according to the judgment of the researcher, if the researcher evaluates that the subject may benefit from the study treatment, they are allowed to be included in the study.
18. Has received a live virus vaccine within 30 days prior to first administration of study drug or plan to be administered during the study period.
19. Known allergy to any component of any investigational drug, known history of severe hypersensitivity to other monoclonal antibody.
20. Known history of mental illness, substance abuse, alcohol, or drug abuse.
21. Is pregnant, breastfeeding women.
22. Any prior or current disease, treatment, or laboratory test abnormality that may confound the study endpoints, interfere with subjects' full participation in the study, or may not be in their best interest to participate in this study.
23. Local or systemic diseases caused by non-malignant tumors, or diseases or symptoms secondary to tumors, which can lead to higher medical risk and/or uncertainty in survival evaluation, such as tumor like leukemia reactions (white blood cell count>20 × 109/L), symptoms of cachexia (known to have lost more than 10% of body weight in the 3 months before screening), etc.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Response Rate (ORR) | from the first drug administration up to two years
  ORR is the proportion of patients with best response of complete response (CR) and partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | from the first drug administration up to two years
  Proportion of patients whose best overall response is either CR, PR, or SD
Duration of response (DOR) | from the first drug administration up to two years
  Time from first documented response (CR or PR) until documented disease progression or death, whichever occurs first
Progression-free Survival (PFS) | from the first drug administration up to two years
  Time from the date of first study treatment administration to the date of first documented tumor progression or death due to any cause, whichever occurs first
Overall survival (OS) | from the first drug administration up to two years
  Time from the date of first study treatment administration to the date of death due to any cause
Adverse event (AE) | From the subject signs the ICF to 90 days after the last dose of study treatment or initiation of other anti-tumor therapy, whichever occurs first
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), and clinically significant abnormal laboratory results

OTHER OUTCOMES:
Biomarkers associated with the response to cadonilimab plus chemotherapy | Samples taken prior to the first dose of drug to confirm the result of MSI-H/dMMR and PD-L1
  Exploration of biomarkers that predict the efficacy of cadonilimab combined with chemotherapy

REFERENCES:
- [Derived] Lin J, Liu T, Chen J, Lin Y, Chen X, Zhuo Y, Li Y, Jiang Y, Yang L, Tu C, Liu B, Zou J, Chen L, Sun Y. Efficacy and safety of cadonilimab combined with chemotherapy as the first-line treatment for primary advanced or recurrent endometrial cancer: a prospective single-arm open-label phase II clinical trial. BMJ Open. 2025 May 19;15(5):e094649. doi: 10.1136/bmjopen-2024-094649. PMID 40389320